CLINICAL TRIAL: NCT01368848
Title: Phase II Study to Investigate the Treatment of Patients With NSCLC Stage IIIB and IV Without the Option of Surgery With a Combination of Cisplatin, Docetaxel and Bevacizumab
Brief Title: Combination of Cisplatin, Docetaxel and Bevacizumab in Patients With Non-small Cell Lung Carcinoma (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Sanofi (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_NSCLC 1; 2008-000765-33 (EudraCT Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: NSCLC
Keywords: AGMT; NSCLC; non-small cell lung cancer; bevacizumab; Avastin; Cisplatin; Docetaxel; Taxotere; Inoperable; stages IIIB and IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab — 3 cycles BCD (Bevacizumab 7,5 mg/kg i.v., Cisplatin 75 mg/m² i.v., Docetaxel 75 mg/m²) Q3W -> Staging
  -> further 3 cycles BCD Q3W -> Bevacizumab Q3W until progression
  Other Names: Avastin
Drug: Cisplatin — 3 cycles BCD (Bevacizumab 7,5 mg/kg i.v., Cisplatin 75 mg/m² i.v., Docetaxel 75 mg/m²) Q3W -> Staging
  -> further 3 cycles BCD Q3W
Drug: Docetaxel — 3 cycles BCD (Bevacizumab 7,5 mg/kg i.v., Cisplatin 75 mg/m² i.v., Docetaxel 75 mg/m²) Q3W -> Staging
  -> further 3 cycles BCD Q3W
  Other Names: Taxotere

SUMMARY:
Despite recent advances in the treatment of NSCLC overall survival within these patients remains dismal and there is yet an unmet medical need for additional treatment options. In this phase II study a combination of chemotherapy with an antibody (cisplatin, docetaxel and bevacizumab) is tested to determine the objective response rate in patients with unresectable and advanced non-small cell lung cancer. This response rate will be compared with historical data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented inoperable, locally advanced, metastatic or recurrent NSCLC other than squamous cell
* At least 1 measurable lesion according to RECIST criteria
* ECOG performance score 0 or 1
* Age between 18 and 70 years

Exclusion Criteria:

* Mixed, non-small cell and small cell tumours or mixed adenosquamous carcinomas with a predominant squamous component.
* History of haemoptysis
* Evidence of tumour invading major blood vessels on imaging.
* Previous neoadjuvant/adjuvant chemotherapy.
* Previous radiotherapy.
* Serious uncontrolled coagulation disorder or thrombo-embolic complications within 6 months prior to study start or history of serious bleeding complications.
* Major surgical procedures within 4 weeks prior to study entry.
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion.
* Non-healing wound, active peptic ulcer or bone fracture.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Response Rate | 4 years
  The primary objective of this proof-of-concept study is to determine the objective response rate in patients with unresectable, stage IIIB and IV non-small cell lung carcinoma treated with the combination cisplatin, docetaxel and bevacizumab. This response rate will be compared to historical data from the ECOG4599 and AVAiL trials.

SECONDARY OUTCOMES:
Progression free survival | 5 years
  Progression free survival, defined as the duration of time from first study treatment until progression or death from any cause as documented by the investigator.
Overall survival | 5 years
  Overall survival, defined as the duration of time from first study treatment until death from any cause.
Duration of response | 5 years
  Duration of response defined as timeframe from first response (CR or PR) until progression from best response.

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Universitaetsklinik der PMU Salzburg, UK f. Innere Medizin III, Salzburg, Salzburg
  - Univ.-Klinik für Innere Medizin V Innsbruck, Abteilung für Hämatologie und Onkologie, Innsbruck, Tyrol
  - Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg